CLINICAL TRIAL: NCT00090168
Title: A Multicenter Study to Assess the Cholesterol Lowering Level of Switching to an Investigational Drug Compared to Doubling the Dose of an Investigational Drug in Patients With Hypercholesterolemia and Atherosclerotic or Coronary Vascular Disease
Brief Title: Cholesterol Lowering Level of MK0653A+Simvastatin in Patients With Hypercholesterolemia and Atherosclerotic or Coronary Vascular Disease (0653A-806)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653A-806; 2004_002
Record Dates: First submitted 2004-08-25; First posted 2004-08-27 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia; Atherosclerotic Disease; Coronary Disease
MeSH Terms: conditions — Hypercholesterolemia; Coronary Disease | interventions — Ezetimibe; Simvastatin; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0653A , ezetimibe (+) simvastatin
Drug: Comparator: atorvastatin
Drug: Duration of Treatment: 6 weeks

SUMMARY:
A 6-week treatment study to compare the reduction in cholesterol of two drugs MK0653A+Simvastatin for high cholesterol, in patients with hypercholesterolemia and atherosclerotic or coronary vascular disease.

ELIGIBILITY:
- Men and women greater than or equal to 18 years of age with elevated cholesterol levels and coronary heart disease (CHD), or atherosclerotic vascular disease may be eligible to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2004-01-27 (Actual); Primary Completion 2004-10-20 (Actual); Study Completion 2004-11-10 (Actual)

PRIMARY OUTCOMES:
LDL-C lowering

SECONDARY OUTCOMES:
Total cholesterol (TC) lowering

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Barrios V, Amabile N, Paganelli F, Chen JW, Allen C, Johnson-Levonas AO, Massaad R, Vandormael K. Lipid-altering efficacy of switching from atorvastatin 10 mg/day to ezetimibe/simvastatin 10/20 mg/day compared to doubling the dose of atorvastatin in hypercholesterolaemic patients with atherosclerosis or coronary heart disease. Int J Clin Pract. 2005 Dec;59(12):1377-86. doi: 10.1111/j.1368-5031.2005.00714.x. PMID 16351668